CLINICAL TRIAL: NCT01959620
Title: Optimal Dose of Early Intervention to Prevent PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Barbara O. Rothbaum, PhD, Professor in Psychiatry and Associate Vice Chair of Clinical Research, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00063758; NARSAD 19798 (Other: Other)
Record Dates: First submitted 2013-10-06; First posted 2013-10-10 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Assessment only (No Intervention): Participants will receive assessment only.
- 1-session exposure intervention (Experimental): Participants will receive one session of exposure therapy.
  Interventions: Behavioral: 1-Session Exposure Therapy
- 3-session exposure intervention (Experimental): Participants will receive three sessions of exposure therapy.
  Interventions: Behavioral: 3-Session Exposure Therapy

INTERVENTIONS:
Behavioral: 1-Session Exposure Therapy — One exposure therapy session lasting one hour
  Arms: 1-session exposure intervention
Behavioral: 3-Session Exposure Therapy — Three exposure therapy sessions lasting one hour each, delivered one week apart
  Arms: 3-session exposure intervention

SUMMARY:
The overall aim of this study is to determine the optimal dose, 3-session exposure intervention versus 1-session exposure intervention compared to no treatment, for the delivery of exposure therapy in the immediate aftermath of trauma for preventing the development of posttraumatic stress disorder.

DETAILED DESCRIPTION:
The precipitant for adult posttraumatic stress disorder (PTSD) is a known event, which allows for immediate intervention and presents the potential to prevent the occurrence of this serious condition. However, there currently are no accepted interventions for the early intervention and prevention of PTSD in the immediate aftermath of trauma. This study will determine whether providing exposure therapy to people who have recently experienced trauma will significantly reduce the severity of PTSD symptoms post-trauma and if delivery of three exposure sessions will result in larger reductions in the symptoms of PTSD post-trauma than one exposure session. This study will also examine predictors for treatment response.

Participation in this study will last 12 months. Participants will first undergo an evaluation session that will include an interview and questionnaires. They will then be randomly assigned to one of the following three conditions: 1-session exposure therapy, 3-session exposure therapy, or assessment only. Participants receiving 1-session exposure therapy will complete one treatment session in the emergency department (ED). Participants receiving 3-session exposure therapy will complete three weekly treatment sessions, with the first occurring in the ED. Treatment will involve reviewing memories of a recent trauma out loud with a therapist and audio-recording these discussions for review at home. All participants will undergo assessments 1, 3, 6, and 12 months after the initial evaluation session.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the emergency department of Emory University School of Medicine/Grady Memorial Hospital for trauma in the past 72 hours
* Meets DSM-IV diagnostic criterion A in which both of the following are present: (i) The person experienced, witnessed, or was confronted with an event or events that involved actual or threatened death or serious injury or a threat to the physical integrity of self or others (ii) The person's response involved intense fear, helplessness, or horror
* Speaks and understands spoken English
* Have a memory of what happened during the trauma
* Can see the assessment forms, hear instructions, and function at an emotional and intellectual level sufficient to allow accurate completion of all assessment instruments

Exclusion Criteria:

* Current or history of mania, schizophrenia, or other psychoses
* Current (past month) prominent suicidal ideation or recent (past 3 months) parasuicidal behavior or other self-injurious behavior, such as low lethality cutting
* Current (past month) substance dependence; people who meet criteria for current substance abuse but not dependence, or past dependence and have been in remission for at least 1 month are eligible
* Experienced a loss of consciousness for more than 5 minutes as a result of injuries sustained during the trauma
* Intoxicated, altered, or highly distressed to the degree that accurate completion of the study assessments or participation in study procedures is not possible
* Blood alcohol level above .08, determined by breathalyzer in the emergency department
* Not alert, oriented, and coherent
* In severe pain, active labor, or respiratory distress or hemodynamically compromised in any way

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Symptom Scale-I (PSS) | Measured 1, 3, 6, 12 months post-trauma

CONTACTS AND LOCATIONS:
Overall Officials: Barbara O. Rothbaum, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Emergency Department, Atlanta, Georgia, United States